CLINICAL TRIAL: NCT06056440
Title: Efficacy of a Physical Rehabilitation Program Using Virtual Reality in Patients With Chronic Tendinopathy (Virtendon-Rehab)
Acronym: VirtendonRehab
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Cadiz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: University of Cadiz PR2022-049; PR2022-049 (Other Grant/Funding Number: University of Cadiz)
Record Dates: First submitted 2023-09-11; First posted 2023-09-28 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2023-09

CONDITIONS: Tendinopathy; Patellar Tendinopathy; Tendinopathy, Elbow; Tendinopathy Rotator Cuff; Achilles Tendinopathy
Keywords: virtual reality; chronic tendinopathy; physical therapy
MeSH Terms: conditions — Tendinopathy; Elbow Tendinopathy | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Outcomes Assessor
Masking Description: A single-blind method will be carried out on the persons collecting and analysing the data
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR group (Experimental): The VR intervention program for the experimental group will be carried through the Oculus Quest 2 device (which consists of VR glasses and different accessories) will be used, in conjunction with software specifically designed for physical rehabilitation of upper and lower limbs: Dynamics VR. This VR intervention will be performed in addition to the patient's usual treatment program.
  Interventions: Procedure: Virtual reality
- Control group (Other)
  Interventions: Other: Control group

INTERVENTIONS:
Procedure: Virtual reality — The VR intervention program for the experimental group will be carried out with a frequency of 3 sessions/week, duration of approximately 45 minutes, and for a total of 12 weeks, being performed in addition to the patient's usual treatment program.
  The Oculus Quest 2 device (which consists of VR glasses and different accessories) will be used, in conjunction with software specifically designed for physical rehabilitation of upper and lower limbs: Dynamics VR. Specifically, the specific functional rehabilitation program will be used, which comprises exercises that are easy to perform, with a playful component, and which encourage the patient's continuous attention to the task performed, acting as a distractor phenomenon in the face of restrictive movement factors such as fear of pain or movement. This software offers the possibility of adjusting the number of repetitions and characteristics of the exercises, thus allowing an individualized physical rehabilitation
  Arms: VR group
Other: Control group — The control group will only receive their usual treatment program for the 12-week duration of the study.
  Arms: Control group

SUMMARY:
Chronic tendinopathies (CT) have a high prevalence (30% of musculoskeletal injuries), causing pain, decreased physical activity and functionality, as well as limitations in daily life. Virtual reality (VR) fosters patient recovery through playful activities that promote competitiveness, stimulates motivation and continuous attention, allows individualizing the exercise program, objectively assessing the execution of the treatment and monitoring the patient's evolution. Therefore, the VIRTENDON-REHAB project aims to conduct a low-risk randomized controlled clinical trial to analyze the efficacy of a VR-based physical rehabilitation program in a population diagnosed with CT on pain, functionality, range of motion, strength, muscle activation pattern, kinesiophobia, quality of life, adherence to treatment and patient satisfaction with the use of the system, compared to a control group. Likewise, the aim is to characterize the clinical profile of this population and to know the relationships between the previous variables. Measurements will be taken at the beginning of the intervention, at the end (12 weeks) and 3 months after the end of the intervention. A descriptive analysis will be performed, inter- and intra-group differences will be analyzed by means of t-Student, Wilcoxon, Mann-Whitney U and mixed ANOVA tests. Cohen's d will be used to determine the effect size. Relationships between variables will be analyzed using structural equations. The results obtained will allow improving knowledge on the management of CT using VR, as well as improving clinical care and reducing healthcare costs.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of tendinopathy (shoulder rotator cuff tendinopathy, epicondylitis/epicondylitis, patellar tendinopathy, achilles tendinopathy).
* Duration of symptoms: greater than 6 weeks.

Exclusion Criteria:

* People who have any pathology that prevents them from performing physical exercise.
* Persons who have undergone surgery.
* Persons who have an illness that may be a contraindication to the proposed procedure.
* Persons who have received exercise therapy in the last 3 months.
* Persons who have received corticosteroid injections in the last 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-11-28 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Disability (Shoulder And Pain Disability Index) | Fom Baseline up to 24 Weeks Follow-up
  Longitudinal change from 0 to 100. Higher scores mean worse outcome.
Disability (Victorian Institute of Sport Assessment - Patellar) | Fom Baseline up to 24 Weeks Follow-up
  Longitudinal change from 0 to 100. Higher scores mean better outcome.
Disability (Victorian Institute of Sport Assessment - Achilles) | Fom Baseline up to 24 Weeks Follow-up
  Longitudinal change from 0 to 100. Higher scores mean better outcome.
Pain (Visual Analogue Scale) | Fom Baseline up to 24 Weeks Follow-up
  Longitudinal change from 0 to 10. Higher scores mean worse outcome.

SECONDARY OUTCOMES:
Range of motion (Goniometer) | Fom Baseline up to 24 Weeks Follow-up
  Longitudinal change
Strength (Dynamometer) | Fom Baseline up to 24 Weeks Follow-up
  Longitudinal change
Kinesiophobia (Tampa Scale Questionnaire) | From Baseline up to 24 Weeks Follow-up
  Longitudinal change from 17 to 68 where the lowest 17 means no or negligible kinesiophobia, and the higher scores indicate an increasing degree of kinesiophobia
Quality of Life (36-item Short Form Survey) | From Baseline up to 24 Weeks Follow-up
  Longitudinal change from 0 to 100. Higher scores mean better outcome.
Adherence (Exercise Adherence Rating Scale) | 12 Weeks and 24 Weeks
  The original English version of the EARS is a 16-item, self-reported questionnaire, which assessadherence of prescribed exercises [6]. The EARS consist of 3 sections. Section 'A' is about prescribedexercise questionnaire. This section consists of 5 questions, which are related to way of doing activitiesand exercise that people often do to improve their physical quality of life. Section 'B' is about exerciseadherence behavior, so called exercise adherence rating scale. This section consists of 6 items, which isan actual measure to identify exercise adherence. This evaluates whether individuals do their exercise asper recommendation or not. Section 'C' is about reasons for adherence/non-adherence of exercises. Thissection consists of 10 items, which assesses factors that hinders and facilitates the exercises. Higher scores mean better outcome.
User satisfaction (Consumer Report Effectiveness Scale) | 12 Weeks and 24 Weeks
  Global satisfaction with the treatment received. 3-item scale scoring from 0 to 300. Higher scores mean better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Nursing and Physiotherapy, Cadiz, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kaux JF, Forthomme B, Goff CL, Crielaard JM, Croisier JL. Current opinions on tendinopathy. J Sports Sci Med. 2011 Jun 1;10(2):238-53. PMID 24149868
- [Background] Mallows A, Debenham J, Walker T, Littlewood C. Association of psychological variables and outcome in tendinopathy: a systematic review. Br J Sports Med. 2017 May;51(9):743-748. doi: 10.1136/bjsports-2016-096154. Epub 2016 Nov 16. PMID 27852585
- [Background] Chen KB, Sesto ME, Ponto K, Leonard J, Mason A, Vanderheiden G, Williams J, Radwin RG. Use of Virtual Reality Feedback for Patients with Chronic Neck Pain and Kinesiophobia. IEEE Trans Neural Syst Rehabil Eng. 2017 Aug;25(8):1240-1248. doi: 10.1109/TNSRE.2016.2621886. Epub 2016 Oct 26. PMID 27810828
- [Background] Dominguez-Tellez P, Moral-Munoz JA, Salazar A, Casado-Fernandez E, Lucena-Anton D. Game-Based Virtual Reality Interventions to Improve Upper Limb Motor Function and Quality of Life After Stroke: Systematic Review and Meta-analysis. Games Health J. 2020 Feb;9(1):1-10. doi: 10.1089/g4h.2019.0043. PMID 32027185
- [Background] Almekinders LC, Almekinders SV. Outcome in the treatment of chronic overuse sports injuries: a retrospective study. J Orthop Sports Phys Ther. 1994 Mar;19(3):157-61. doi: 10.2519/jospt.1994.19.3.157. PMID 8156067
- [Background] Cook JL, Purdam CR. Is tendon pathology a continuum? A pathology model to explain the clinical presentation of load-induced tendinopathy. Br J Sports Med. 2009 Jun;43(6):409-16. doi: 10.1136/bjsm.2008.051193. Epub 2008 Sep 23. PMID 18812414
- [Derived] Lucena-Anton D, Dominguez-Romero JG, Chacon-Barba JC, Santi-Cano MJ, Luque-Moreno C, Moral-Munoz JA. Efficacy of a physical rehabilitation program using virtual reality in patients with chronic tendinopathy: A randomized controlled trial protocol (VirTendon-Rehab). Digit Health. 2025 Feb 18;11:20552076241297043. doi: 10.1177/20552076241297043. eCollection 2025 Jan-Dec. PMID 39974760
- See also: Virtual reality software — https://www.dynamics-vr.com